CLINICAL TRIAL: NCT00158080
Title: Prevention of Contrast-Induced Nephropathy by Real-Time Hemofiltration
Brief Title: Hemofiltration for Contrast-Induced Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nara Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K0001
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Kidney Disease; Cardiac Catheterization
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Hemofiltration

INTERVENTIONS:
Procedure: hemofiltration

SUMMARY:
Contrast-induced acute renal failure can be prevented with hemofiltration which is performed during cardiac catheterization

ELIGIBILITY:
Inclusion Criteria:

* Patients with serum creatinine>2.0mg/dl and/or GFR<50ml/min

Exclusion Criteria:

* Emergent cardiac catheterization
* Patients on chronic dialysis
* Patients with HYHA>III heart failure

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

PRIMARY OUTCOMES:
Prevention of contrast-induced acute renal failure, Elevation of serum creatinine

SECONDARY OUTCOMES:
Need for hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiko Saito, MD, PhD, Study Director — Nara Medical University
Locations (1):
- First Dept of InternalMedicine, Nara Medical University, Kashihara, Nara, Japan

REFERENCES:
- [Background] Kashyap AS, Anand KP, Kashyap S. Hemofiltration and the prevention of radiocontrast-agent-induced nephropathy. N Engl J Med. 2004 Feb 19;350(8):836-8; author reply 836-8. No abstract available. PMID 14978842